CLINICAL TRIAL: NCT06123468
Title: A Phase Ib/II Single-arm, Multicenter Study of Sacituzumab-govitecan, a TROP-2 Targeting Antibody Linked With SN38, for Patients With Metastatic Esophagogastric Adenocarcinoma
Brief Title: Study Evaluating Treatment of Sacituzumab-govitecan for Patients With Metastatic Esophagogastric Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAGA; 2023-505257-40-00 (Other: EU CT Number); AIO-STO-0123/ass. (Other: AIO); IKF-t065 (Other: IKF Trial ID)
Record Dates: First submitted 2023-11-06; First posted 2023-11-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: gastric adenocarcinoma; GEJ adenocarcinoma
MeSH Terms: interventions — sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: All eligible enrolled patients will receive Sacituzumab-govitecan 10 mg/kg i.v. at day 1 and day 8 of each 21-day cycle (Q3W).
  Patients will receive the treatment for a maximum of 12 months or until disease progression, unacceptable toxicity or withdrawal of consent, whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab-govitecan (Experimental): Single arm with Sacituzumab-govitecan 10 mg/kg i.v. at day 1 and day 8 of each 21-day cycle (Q3W). Patients will receive the treatment for a maximum of 12 months.
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — 10 mg/kg i.v. at day 1 and day 8 of each 21-day cycle (Q3W) for max 17 cycles (max. 12 months treatment)
  Other Names: Trodelvy

SUMMARY:
The study is a open-label, single-arm, multicenter, phase Ib/II trial assessing the efficacy of sacituzumab-govitecan for metastatic esophagogastric adenocarcinoma

DETAILED DESCRIPTION:
All eligible enrolled patients will receive:Sacituzumab-govitecan 10 mg/kg i.v. at day 1 and day 8 of each 21-day cycle (Q3W). Patients will receive the treatment for a maximum of 12 months or until disease progression, unacceptable toxicity or withdrawal of consent, whichever occurs first.The primary objective of the trial is to evaluate the efficacy (primary endpoint: Overall Response Rate ORR, complete response + partial response) of sacituzumab-govitecan for metastatic esophagogastric adenocarcinoma. The secondary objectives are to further characterize the efficacy of sacituzumab-govitecan for metastatic esophagogastric adenocarcinoma and to evaluate safety and tolerability of sacituzumab-govitecan for metastatic esophagogastric adenocarcinoma. Secondary endpoints comprise the assessment of Clinical benefit rate (CBR, complete response + partial response + stable disease), Progression-free survival (PFS), Overall survival (OS), ORR, CBR, PFS and OS in the subgroup of TROP-2 overexpression, toxiticy. In addition, tissue and blood samples will be analyzed to evaluate the TROP-2 expression during treatment with sacituzumab-govitecan for metastatic esophagogastric adenocarcinoma.

56 patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* has given written informed consent.
2. Patient is, in the investigator's judgement, willing and able to comply with the study protocol.
3. Patient is ≥ 18 years of age at time of signing the written informed consent.
4. Patient has been diagnosed with histologically confirmed metastatic (stage IV) esophagogastric adenocarcinoma.
5. Patient has received at least one prior therapy containing platinum compound and a fluoropyrimidine, potentially combined with immunotherapy, in the metastatic setting. Neoadjuvant/adjuvant platinum-fluoropyrimidine treatment is counted as first-line therapy if disease progression occurred within 6 months after completion of treatment.

   NOTE: patients with advanced MSI-h/dMMR tumors who have not previously been treated with pembrolizumab, nivolumab or any other PD-1/PD-L1 inhibitor are not permitted for inclusion.
6. Patient has an ECOG performance status ≤ 1.
7. Patient must have an estimated life expectancy of at least 12 weeks.
8. Patient has at least one measurable lesion on radiographic imaging as defined by RECIST v1.1.
9. Patient has adequate hematological, hepatic and renal function as indicated by the following parameters:

   1. Leukocytes ≥ 2,500/μL, platelets ≥ 100,000/μL without transfusion, absolute neutrophil count (ANC) ≥ 1,500/μL without granulocyte colony-stimulating factor support, hemoglobin ≥ 90 g/L (9 g/dL) - Patients may be transfused to meet this criterion.
   2. Bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate transaminase and alanine transaminase ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastases), alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastases)
   3. Serum creatinine ≤ 1.5 x ULN, or glomerular filtration rate > 45 mL/min (calculated per institutional standard)
   4. Serum albumin ≥ 25 g/L (2.5 g/dL)
   5. For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN; for patients receiving therapeutic anticoagulation: stable anticoagulant regimen
10. Patient must be willing to provide liquid biopsy samples for the translational research program.
11. Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last study treatment. Male patients must refrain from donating sperm during this same period. Male patients with a pregnant partner must agree to

Exclusion Criteria:

1. Patient has known hypersensitivity to any component of the Sacituzumab-govitecan formulation as well as a known history of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
2. Patient has received previously topoisomerase 1 inhibitors such as irinotecan, or nal-irinotecan
3. Patient has an active second malignancy. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (e.g., non-melanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll
4. Patients with known, untreated and active (not stable within the last 4 weeks or symptomatic) brain metastases and patients with leptomeningeal disease.
5. Patient meets any of the following criteria for cardiac disease:

   1. Myocardial infarction or unstable angina pectoris within 6 months prior to initiation of study treatment
   2. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular bock, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
   3. New York Heart Associated (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction (LVEF) of < 40% if echocardiography has been performed
6. Patient has an active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months prior to initiation of study treatment
7. Patient has an active serious infection requiring antibiotic treatment
8. Patient has known history of human immune deficiency virus (HIV, or positive HIV antibody, if done at screening) with detectable viral load OR taking medications that may interfere with SN-38 metabolism
9. Patient has active hepatitis B or C virus (HBV/HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded
10. Patient participated in another interventional clinical study ≤ 14 days prior to initiation of study treatment or at the same time as this study.
11. Patient has taken an investigational drug within 14 days or 5 half-lives (whichever is longer) prior to initiation of study treatment.
12. Patient received anticancer biologic agent within 28 days or targeted small molecule, radiation or chemotherapy within 14 days prior to initiation of the study treatment.
13. Patient has not recovered from AEs due to previously administered drug (i.e., ≥ grade 2 is concerned as not recovered)

    1. Patients with any grade of alopecia are an exception to this criterion and will qualify for the study
    2. If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
14. Patient has evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results.
15. Female patients, who are pregnant or breast feeding or planning to become pregnant within and 6 months after the end of treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | up to 12 months
  Objective response rate will be assessed according to RECIST v1.1. criteria and is defined as proportion of patients showing complete or partial response (CR+PR).

SECONDARY OUTCOMES:
Clinical benefit rate | up to 36 months
  Clinical benefit rate will be assessed according to RECIST v1.1. criteria and is defined as proportion of patients showing complete response, partial response or stable disease (CR+PR+SD).
Progression-free survival (PFS) | up to 36 months
  Progression-free survival is defined as time from enrollment to the date of progression according to RECIST v1.1 or death due to any cause. Patients who have not experienced an event at the time of analysis will be censored at the most recent date of disease assessment.
Overall survival (OS) | up to 36 months
  Overall survival is defined as the time from enrollment to the date of death from any cause. Patients who have not experienced an event at the time of analysis will be censored at the date when the patient was last known to be alive.
Safety and toxicity | up to 13 months (max. 12 months treatment plus 30 days after last treatment)
  Safety and tolerability assessments will include physical examinations, clinical laboratory profile and continuous assessments of adverse events (AEs).
  AEs will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (8):
- SCRI-CCCIT GmbH, Salzburg, Austria
- Germany (7):
  - Hämatologisch-Onkologische Praxis Eppendorf, Hamburg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Onkopraxis Probstheida, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar der TU München, München

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Kobitzsch B, Stocker G, Hacker UT, Junge S, Pauligk C, Al-Batran SE, Goetze TO, Lordick F. SAGA-a phase Ib/II single-arm, multicenter study of sacituzumab govitecan for patients with metastatic esophagogastric adenocarcinoma. ESMO Gastrointest Oncol. 2024 Apr 12;4:100051. doi: 10.1016/j.esmogo.2024.100051. eCollection 2024 Jun. PMID 41648033